CLINICAL TRIAL: NCT06453889
Title: Efficacy and Safety of Multimode Thermal Therapy in the Treatment of Early Peripheral Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KS24015
Record Dates: First submitted 2024-05-25; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: multimode thermal therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimode thermal therapy (Experimental): Percutaneous multimode thermal therapy
  Interventions: Device: Multimode thermal therapy

INTERVENTIONS:
Device: Multimode thermal therapy — The multimode thermal therapy procedure consists of a sequential rapid freezing, natural thawing, and radio-frequency (RF) heating of the target tumor tissue.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of multimode thermal therapy for early peripheral lung cancer, and to explore the changes of systemic immune microenvironment after multimode thermal therapy.

DETAILED DESCRIPTION:
This is a single-center, single-arm, exploratory study, and is expected to enroll a total of 10 patients. The enrolled patients were stage IA lung cancer patients with lung lesions found on chest CT, pathologically diagnosed as non-small cell lung cancer, negative for driver gene mutations, and who were considered high-risk or refused surgery by multidisciplinary evaluation. Follow-ups are performed after the multimode thermal therapy. The primary endpoint is complete ablation rate at 6 months after multimode thermal therapy. The secondary endpoints are complete ablation rate at 12 months after multimode thermal therapy, local control rate at 1, 2, 3 years post-procedure, progression-free survival and mmune effects after multimodal thermal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Pathologically diagnosed as primary peripheral non-small cell lung cancer, preoperative staging suggested clinical staging as T1N0M0, stage IA (including new-onset lung cancer after surgery and multiple primary lung cancer);
3. The ECOG PS score is 0-2;
4. Expected survival ≥6 months;
5. Negative driver gene mutation: driver genes were defined as EGFR, ALK, ROS1, RET;
6. Agree to undergo multimode thermal therapy as initial treatment after being assessed unsuitable for surgery or refusing surgery, and sign informed consent.

Exclusion Criteria:

1. Patients with poor cardiopulmonary function or other comorbidities who cannot tolerate multimode thermal therapy;
2. Patients whose chest CT indicated that the lung lesions could not be reached through the chest wall through multimode thermal therapy;
3. Severe liver and kidney function and coagulation function abnormalities, platelet count <70×109/L;
4. Poor control of malignant pleural effusion;
5. Patients who have received other anti-tumor drugs or have used immune checkpoint inhibitors in the past 6 months;
6. The patient has an uncontrolled disease (including but not limited to active infection, symptomatic congestive heart failure, unstable angina, arrhythmia, mental illness, etc.);
7. Those who have undergone surgical operations or had allogeneic organ transplants within 1 month;
8. Primary immune deficiency or autoimmune diseases (e.g. rheumatoid arthritis, systemic lupus erythematosus, etc.);
9. Pregnant and lactating women;
10. Long-term use of steroid;
11. Other circumstances considered inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-05 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate at 6 months post-procedure | 6 months
  This refers to the proportion of completely ablated lesions in the total ablated lesions at 6 months after multimode thermal therapy.

SECONDARY OUTCOMES:
Complete ablation rate at 12 months post-procedure | 12 months
  This refers to the proportion of completely ablated lesions in the total ablated lesions at 12 months after multimode thermal therapy.
Local control rate at 1, 2, 3 years post-procedure | 3 years
  This refers to the proportion of completely and incompletely ablated lesions in the total ablated lesions at 1 year, 2 years and 3 years after multimode thermal therapy.
Progression-free survival | 3 years
  This refers to the length of time between the participant's first onset of disease progression or death from any cause after multimode thermal therapy.
Immunological response (lymphocyte phenotypes, PD-L1 expression, cytokines) | 3 months
  This refers to the changes from baseline in the immunological responses following the multimode thermal therapy, including the percentage and function of lymphocyte phenotypes, the expression of PD-L1, the concentration of IL-6/IL-17A levels, etc.
Number of participants with adverse events | 1 month
  This refers to all treatment-related adverse events (grade 1- 5) occurring during the trial and follow-up period as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No